CLINICAL TRIAL: NCT05857852
Title: Low-Intensity Focused Ultrasound for Cocaine Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Professor of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HSR220247
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Cocaine Use Disorder; Cocaine Dependence; Cocaine Abuse; Ultrasound
Keywords: Substance Use Disorders; Chemically-Induced Disorders; Substance-related disorders; Cocaine Addiction; Cocaine
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders

STUDY DESIGN:
Intervention Model Description: At each of two intervention visits, participants will receive either LIFU or sham. At the completion of both visits, all participants will have received both, LIFU and sham.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Low-Intensity Focused Ultrasound (LIFU) (Experimental): All subjects to receive LIFU and Sham in a randomized order.
  Interventions: Device: Low-Intensity Focused Ultrasound
- Sham LIFU (Sham Comparator): All subjects to receive LIFU and Sham in a randomized order.
  Interventions: Device: Sham LIFU device

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound — Low-Intensity Focused Ultrasound administration to right dorsal anterior insula, in one of two sessions
  Arms: Low-Intensity Focused Ultrasound (LIFU)
Device: Sham LIFU device — Sham LIFU device administered in one of two sessions
  Arms: Sham LIFU

SUMMARY:
This study aims to understand the role of Low-Intensity Focused Ultrasound on craving levels for cocaine as evidenced by diagnostic imaging of the dorsal anterior insula (dAI) and subjective ratings. Data analysis will serve to show if 1) LIFU is safe and effective and to 2) examine the effects of LIFU on dAI BOLD activity and craving in response to cocaine cue-exposure. The study will screen 60 individuals with Cocaine Use Disorder (CUD) to arrive at 30 enrolled subjects, based on a 2:1 screen/randomization ratio.

DETAILED DESCRIPTION:
This is a randomized single-blind, active, sham-controlled study.

This study will enroll thirty (30) individuals, aged 18 years and older, that meet the criteria for CUD. Participants will be recruited from the general population and will be asked to complete cognitive testing and measures, self-reported craving measures, and diagnostic exams including magnetic resonance imaging (MRI) and Computed Tomography (CT). Participants will also undergo functional MRI which entails being shown cocaine-related photos at regular intervals.

All participants will receive LIFU and sham interventions, but will be randomized to one of two sessions, and will return one month after the second session for an in-person follow-up. In total, there are five (5) in-person visits and two (2) phone calls to assess for adverse events, conducted over eight (8) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older with a history of cocaine use disorder
* Have a current (past 6 months) DSM-5 diagnosis of cocaine use disorder (4 or more symptoms) assessed using the MINI neuropsychiatric interview
* Have a blood alcohol content by breathalyzer, equal to 0.000 when informed consent document is signed
* Ability to abstain from cocaine use at key points during study
* Willingness and ability to comply with scheduled visits and study procedures
* Ability to lie down for extended periods of time for imaging tests
* Will have reliable transportation throughout study
* Will have a stable residence during the 2 weeks prior to randomization and not be at risk of losing housing in next 2 months
* Must meet criteria to have magnetic resonance imaging (MRI)

Exclusion Criteria:

• Please contact PI or Study Coordinator for more details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in Bold Oxygen Level Dependent (BOLD)% signal change in response to cocaine cue exposure | 8 weeks
  Evidence on MRI of BOLD activity in the dAI region
Decrease in average craving score by 25% for LIFU compared to sham | 8 weeks
  Participant, subjective rating of cocaine-related craving
No evidence of neurological or other adverse events related to LIFU | 8 weeks
  MRI images will show congruity of brain data over course of study

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, MD, Principal Investigator — University of Virginia, Center for Leading Edge Addiction Research
Locations (1):
- UVA Center for Leading Edge Addiction Research, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No